CLINICAL TRIAL: NCT04870138
Title: Experimental Human Infection With Isogenic Mutants of Neisseria Gonorrhoeae (LptA Trial)
Brief Title: Experimental Human Infection With Neisseria Gonorrhoeae (LptA Trial)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0106 LptA
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2020-09

CONDITIONS: Gonococcal Infection
Keywords: ceftriaxone; challenge; ciprofloxacin; males; Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — Azithromycin; Ceftriaxone; Ciprofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mixed FA7527/FA1090 (Experimental): Bacterial inoculum containing a mixture of equivalent numbers of the isogenic LptA mutant and wild-type (WT) strain administered once to the anterior urethra. N= up to 25
  Interventions: Drug: Azithromycin; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA1090 A26; Biological: Neisseria gonorrhoeae strain FA7527
- Mutant FA7527 (Experimental): Bacterial inoculum containing only the isogenic LptA mutant N. gonorrhoeae strain administered once to the anterior urethra. N= up to 8
  Interventions: Drug: Azithromycin; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA7527
- Wild-type FA1090 (Experimental): Bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain administered once to the anterior urethra. N= up to 8
  Interventions: Drug: Azithromycin; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA1090 A26

INTERVENTIONS:
Drug: Azithromycin — Alternative antibiotic treatment failure therapy: Azithromycin 2 g orally in a single dose after treatment failure with both cephalosporin and quinolone antibiotics.
Drug: Ceftriaxone — Mandatory antibiotic treatment failure therapy: Ceftriaxone 250 mg intramuscular in a single dose on patient request, at the onset of symptoms, or on the 5th study day after inoculation.
Drug: Ciprofloxacin — Mandatory antibiotic treatment failure therapy: Ciprofloxacin 500 mg orally in a single dose on patient request, at the onset of symptoms or on the 5th study day after inoculation.
Biological: Neisseria gonorrhoeae strain FA1090 A26 — 0.4 mL of a suspension containing 10^5 - 10^6 CFU of wild-type (WT) Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
  Arms: Mixed FA7527/FA1090; Wild-type FA1090
Biological: Neisseria gonorrhoeae strain FA7527 — 0.4 mL of a suspension containing 10^5 - 10^6 CFU of isogenic LptA mutant Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
  Arms: Mixed FA7527/FA1090; Mutant FA7527

SUMMARY:
This is a Phase 1, interventional, non-randomized, experimental infection model study in healthy adult males (N=up to 25) between the ages of 18-35 at study enrollment. The study is designed to test the requirements of predicted N. gonorrhoeae virulence determinants for gonococcal infection in the male urethra through infection with engineered mutants of N. gonorrhoeae. We predict that mutations abolishing expression of N. gonorrhoeae virulence determinants will eliminate or significantly reduce gonococcal infectivity or the ability to induce inflammation in an infected individual, thus identifying potential vaccine candidates. Study duration will be 1 year, and the duration for all participants will be about 3 weeks. The primary objective of the study is to compare the ability of different engineered mutants of Neisseria gonorrhoeae to cause a clinical infection (signs or symptoms of urethritis such as discomfort during urination, urethral discharge, etc.) in the male urethra.

DETAILED DESCRIPTION:
This is a Phase 1, interventional, non-randomized, experimental infection model study in healthy adult males (N=up to 25) between the ages of 18-35 at study enrollment. The study is designed to test the requirements of predicted N. gonorrhoeae virulence determinants for gonococcal infection in the male urethra through infection with engineered mutants of N. gonorrhoeae. We hypothesize that key virulence determinants involved in N. gonorrhoeae adherence and resistance to innate immunity are essential for infection in the male urethra. We predict that mutations abolishing expression of these virulence determinants will eliminate or significantly reduce gonococcal infectivity or the ability to induce inflammation in an infected individual, thus identifying potential vaccine candidates. For each mutant to be investigated under this protocol, initial trials will be conducted in which subjects receive a bacterial inoculum containing a mixture of equivalent numbers of two isogenic strains, differing in expression of one or more genes. A competitive advantage for one strain during urethral infection will be manifest by recovery of that strain in a statistically significantly higher proportion of isolates recovered from infected subjects than in the inoculum. Following infections with mixed inocula, infectivity of the mutant in single-strain infections will be compared to that of the wild-type in single-strain infections. In addition, the proportion of infected subjects that develop signs or symptoms of urethritis with mutant and wild- type inocula will be compared. The Mixed FA7527/FA1090 group (n = up to 25 ) will receive a bacterial inoculum containing a mixture of equivalent numbers of the isogenic mutant and WT strains. In single-strain infections, the Mutant FA7527 group (n = up to 8) will receive a bacterial inoculum containing only the isogenic mutant N. gonorrhoeae strain, and the Wild-type FA1090 group (n = up to 8) will receive a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain. All subjects will be examined daily for symptoms of infection and receive antibiotic treatment at the end of the inpatient portion of the trial. Study duration will be 1 year, and the duration for all participants will be about 3 weeks. The primary objective of the study is to compare the ability of different engineered mutants of Neisseria gonorrhoeae to cause a clinical infection (signs or symptoms of urethritis such as discomfort during urination, urethral discharge, etc.) in the male urethra. The study secondary objectives are to: (1) characterize host immune responses to infection by measuring cytokines and other mediators in specimens including serum, peripheral blood lymphocytes and urine obtained from subjects before, during and after experimental gonococcal infection, and (2) characterize bacterial gene expression during experimental infection.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man between the ages of 18 and 35 years.
2. Able and willing to be located easily by providing street address and telephone number (land line and/or cell phone number).
3. Willingness to provide written informed consent.
4. Able and willing to attend all study visits including 6-day stay in the Clinical and Translational Research Center (CTRC) during the trial (with ability to leave the unit during the day) and follow-up visit during the week after treatment.
5. Able and willing to abstain from masturbation during the 6-day stay in the CTRC.
6. Able and willing to abstain from all sexual activity during the course of the study.
7. Acceptable medical history by screening evaluation.
8. Standard physical exam within normal limits (WNL).
9. Serum creatinine WNL.
10. Serum alanine transaminase (ALT) WNL.
11. White blood cell (WBC), polymorphonuclear cell (PMN) and hemoglobin values WNL.
12. Normal urinalysis.
13. Total Complement (CH50) WNL.
14. Urine negative for chlamydia, gonorrhea, trichomonas and mycoplasma.
15. Negative HIV, syphilis, and Hepatitis C (HCV) test results.
16. Negative Hepatitis B (HBV) core and surface antibodies or results consistent with immunization (negative HBV core antibody/positive HBV surface antibody).
17. Denies history of STIs including syphilis and hepatitis B & C.
18. Denies history of bleeding diathesis.
19. Denies history of seizures (due to reports of seizures with ciprofloxacin).
20. Denies history of cancer, except basal cell carcinoma of the skin more than 5 years ago.
21. Denies history of drug abuse.
22. Denies history of psychiatric disorders, except depression controlled by medication.
23. Denies history of genitourinary surgery.

Exclusion Criteria:

1. Student or employee under the direct supervision of any of the study investigators.
2. Any known immunodeficiencies including complement deficiency, antibody deficiency, chronic granulomatous disease or HIV infection.
3. Psychiatric disorders that would interfere with the integrity of the data or volunteer safety.
4. Unstable depression (defined as receiving either < 3 months of the same medication (and dose) or a decompensating event during the previous 3 months) or depression that, in the opinion of the investigator, will compromise the subject's ability to comply with protocol requirements.
5. Heart murmur or heart disease.
6. Anatomic abnormality of the urinary tract.
7. Any antibiotic treatment in the past 30 days, or azithromycin in the past 60 days.
8. Chemotherapy within the past year.
9. Current steroid use, except for topical application.
10. Allergy to penicillin, ceftriaxone or ciprofloxacin or to lidocaine.
11. Treatment with medications that are contraindicated with ciprofloxacin or ceftriaxone and that cannot be withheld for the single doses given in this study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03-10 (Actual); Primary Completion 2015-04-28 (Actual); Study Completion 2015-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina Health Care - Infectious Diseases, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males aged 18-<36 years old, living in central North Carolina, in general good health with no history of sexually transmitted infections (STIs) were enrolled. Participants were enrolled between 10MAR2013 and 26APR2015.
Groups:
- Mutant FA7527 - LptA: Participants received a bacterial inoculum containing only the isogenic LptA mutant N. gonorrhoeae strain.
  Neisseria gonorrhoeae strain FA7527: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter. Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose; or Ciprofloxacin 500 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
- Wild-type FA1090 A25: Participants received a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain.
  Neisseria gonorrhoeae strain FA1090 A25: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter. Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose; or Ciprofloxacin 500 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
- Mixed FA7527/FA1090 A25: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic LptA mutant and WT strain.
  Neisseria gonorrhoeae strains FA7527 and FA1090 A25: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter. Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose; or Ciprofloxacin 500 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
Period: Overall Study
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25 | Mixed FA7527/FA1090 A25
Started | 5 | 5 | 6
Completed | 5 | 5 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants.
Groups:
- Mutant FA7527 - LptA: Participants received a bacterial inoculum containing only the isogenic LptA mutant N. gonorrhoeae strain. Mandatory rescue therapy in a single dose, on participant request, at the onset of symptoms or on the 5th study day after inoculation.
- Wild-type FA1090: Participants received a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain. Mandatory rescue therapy in a single dose, on participant request, at the onset of symptoms or on the 5th study day after inoculation.
- Mixed FA7527/FA1090: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic LptA mutant and WT strain. Mandatory rescue therapy in a single dose, on participant request, at the onset of symptoms or on the 5th study day after inoculation.
- Total: Total of all reporting groups
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 | Mixed FA7527/FA1090 | Total
Number analyzed (Participants) | 5 | 5 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.3 (2.6) | 22.1 (2.3) | 24.9 (3.3) | 23.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 5 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 5 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 2 | 4 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants That Become Infected With Individual N. Gonorrhoeae Strains in Non-competitive Infections
Description: Infection defined as reported symptoms of urethritis, including urethral discharge or dysuria, plus presence of gram-negative intracellular diplococci in a urethral swab smear. The proportion of infected participants by Day 5 with N. gonorrhoeae was assessed by group among participants with non-competitive infections. Participants could become infected and received treatment any day before or on day 5.
Time Frame: Day of infection, any day between Day 1 and Day 5
Population: All participants inoculated with a dose of N. gonorrhoeae within 1 log10 of the intended dose and reached an objective study endpoint (symptoms of urethritis or day 5)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Wild-type FA1090 A25: Participants received a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain. Mandatory rescue therapy in a single dose, on participant request, at the onset of symptoms or on the 5th study day after inoculation.
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
proportion of participants | 0.80 [0.28 to 0.99] | 1.00 [0.47 to 1.00]
Statistical Analysis 1: Comparison: Mutant FA7527 - LptA vs Wild-type FA1090 A25; Test type: Other; p = 1.000, Fisher Exact — One-sided Fisher's Exact Test with alpha = 0.05

2. Primary Outcome: The Proportion of Participants That Become Infected With Mixed Inoculum
Description: Infection defined as reported symptoms of urethritis, including urethral discharge or dysuria, plus presence of gram-negative intracellular diplococci in a urethral swab smear. Participants could become infected and received treatment any day before or on day 5.
Time Frame: Day of infection, any day between Day 1 and Day 5
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Mixed FA7527/FA1090 A25: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic LptA mutant and WT strain. Mandatory rescue therapy in a single dose, on participant request, at the onset of symptoms or on the 5th study day after inoculation.
Arm/Group | Mixed FA7527/FA1090 A25
Number analyzed (Participants) | 6
proportion of participants | 0.83 [0.36 to 1.00]

3. Primary Outcome: The Proportion of Wild Type (WT) Organisms Recovered From Urine and Urethral Swab Specimens From Individual Subjects Infected With Mixed Inoculum
Description: as for outcome 2
Time Frame: Baseline (Day 0) and the day of infection (any day between Day 1 and Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of WT organisms recovered
Groups:
- Mixed FA7527/FA1090 A25: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic LptA mutant and WT strain. Mandatory rescue therapy in a single dose, on patient request, at the onset of symptoms or on the 5th study day after inoculation.
Arm/Group | Mixed FA7527/FA1090 A25
Number analyzed (Participants) | 5
proportion of WT organisms recovered | 1.0 (0.0)
Statistical Analysis 1: Comparison: Mixed FA7527/FA1090 A25; Null hypothesis: The proportion of the strain in the inoculum = 0.5; Test type: Other; p < 0.0001, t-test, 1 sided; One-sided single sample t-test with alpha=0.05

4. Secondary Outcome: EGF Cytokine Levels in Peripheral Blood
Description: EGF Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: Screening Visit (Day -30 to Day -1), Treatment Visit (Day 1 to Day 5), and Follow-Up Visit (3 to 7 days following Treatment Visit)
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with EGF Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 85.0 [1.8 to 189.6] | 33.5 [1.8 to 82.6]
  Treatment Visit | 42.6 [2.9 to 82.3] | 29.6 [1.8 to 73.1]
  Follow-Up Visit | 37.9 [1.8 to 79.2] | 42.9 [1.8 to 92.5]

5. Secondary Outcome: Eotaxin Cytokine Levels in Peripheral Blood
Description: Eotaxin cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with Eotaxin Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 351.9 [91.6 to 612.2] | 267.4 [162.9 to 371.9]
  Treatment Visit | 422.7 [25.7 to 819.7] | 247.3 [25.9 to 468.7]
  Follow-Up Visit | 407.1 [1.5 to 840.8] | 218.3 [69.5 to 367.1]

6. Secondary Outcome: G-CSF Cytokine Levels in Peripheral Blood
Description: G-CSF Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with G-CSF Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 32.5 [1.8 to 74.5] | 81.6 [1.8 to 258.7]
  Treatment Visit | 37.8 [8.5 to 67.1] | 91.4 [1.8 to 293.1]
  Follow-Up Visit | 19.2 [1.8 to 54.5] | 72.9 [1.8 to 207.7]

7. Secondary Outcome: Fractalkine Cytokine Levels in Peripheral Blood
Description: Fractalkine Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with Fractalkine Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 202.2 [43.5 to 440.0] | 761.8 [43.5 to 1912.4]
  Treatment Visit | 248.3 [43.5 to 512.6] | 762.9 [43.5 to 1989.2]
  Follow-Up Visit | 222.2 [43.5 to 471.4] | 853.7 [43.5 to 2234.9]

8. Secondary Outcome: GRO Cytokine Levels in Peripheral Blood
Description: GRO Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with GRO Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 1003.9 [297.2 to 1710.6] | 433.5 [63.9 to 803.1]
  Treatment Visit | 436.4 [253.7 to 619.1] | 507.3 [297.0 to 717.6]
  Follow-Up Visit | 403.1 [201.4 to 604.8] | 605.5 [354.4 to 856.6]

9. Secondary Outcome: IL-1RA Cytokine Levels in Peripheral Blood
Description: IL-1RA Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with IL-1RA Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 145.6 [1.9 to 446.0] | 104.5 [1.9 to 319.4]
  Treatment Visit | 144.0 [1.9 to 401.4] | 94.0 [1.9 to 277.2]
  Follow-Up Visit | 106.2 [1.9 to 293.6] | 97.7 [1.9 to 289.1]

10. Secondary Outcome: IL-8 Cytokine Levels in Peripheral Blood
Description: IL-8 Cytokine levels in peripheral blood collected from subjects were measured at the eligibility testing visit, during experimental infection and at the follow-up visit. Only cytokines detected during experimental infection in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with IL-8 Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 17.3 [1.6 to 37.7] | 22.1 [1.6 to 67.3]
  Treatment Visit | 23.0 [5.5 to 40.5] | 21.6 [1.6 to 66.2]
  Follow-Up Visit | 18.0 [1.6 to 37.4] | 21.2 [1.6 to 62.7]

11. Secondary Outcome: IP-10 Cytokine Levels in Peripheral Blood
Description: IP-10 Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with IP-10 Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 630.8 [200.2 to 1061.4] | 598.4 [1.7 to 1212.6]
  Treatment Visit | 781.0 [549.0 to 1013.0] | 790.3 [37.9 to 1542.7]
  Follow-Up Visit | 516.0 [338.2 to 693.8] | 361.9 [103.9 to 619.9]

12. Secondary Outcome: MCP-1 Cytokine Levels in Peripheral Blood
Description: MCP-1 Cytokine levels in peripheral blood collected from subjects were measured at the eligibility testing visit, during experimental infection and at the follow-up visit. Only cytokines detected during experimental infection in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with MCP-10 Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 428.0 [216.0 to 640.0] | 339.7 [181.5 to 497.9]
  Treatment Visit | 563.0 [434.7 to 691.3] | 271.7 [199.4 to 344.0]
  Follow-Up Visit | 379.2 [219.7 to 538.7] | 284.1 [168.3 to 399.9]

13. Secondary Outcome: MIP-1Beta Cytokine Levels in Peripheral Blood
Description: MIP-1Beta Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with MIP-1Beta Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 45.4 [1.3 to 95.4] | 42.9 [1.3 to 139.2]
  Treatment Visit | 48.4 [9.2 to 87.6] | 37.8 [1.3 to 127.9]
  Follow-Up Visit | 39.4 [1.3 to 82.0] | 36.0 [1.3 to 122.0]

14. Secondary Outcome: VEGF Cytokine Levels in Peripheral Blood
Description: VEGF Cytokine levels in peripheral blood collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with VEGF Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 321.1 [44.0 to 744.5] | 480.7 [44.0 to 1466.2]
  Treatment Visit | 340.3 [44.0 to 706.8] | 376.7 [44.0 to 1235.9]
  Follow-Up Visit | 334.1 [44.0 to 745.3] | 409.9 [44.0 to 1310.9]

15. Secondary Outcome: EGF Cytokine Levels in Urine
Description: EGF Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 7333.2 [4942.2 to 8525.2] | 6600.9 [3086.1 to 8525.2]
  Treatment Visit | 7358.1 [4270.2 to 8525.2] | 8325.2 [7786.5 to 8525.2]
  Follow-Up Visit | 7358.1 [4270.2 to 8525.2] | 8490.4 [8393.5 to 8525.2]

16. Secondary Outcome: Eotaxin Cytokine Levels in Urine
Description: Eotaxin Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 5.2 [1.7 to 37.7] | 2.7 [1.0 to 4.4]
  Treatment Visit | 5.9 [1.7 to 10.6] | 5.4 [1.7 to 11.0]
  Follow-Up Visit | 7.1 [1.7 to 13.9] | 2.2 [1.7 to 3.5]

17. Secondary Outcome: G-CSF Cytokine Levels in Urine
Description: G-CSF Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 16.6 [3.3 to 29.9] | 25.6 [1.5 to 64.4]
  Treatment Visit | 113.1 [16.5 to 209.7] | 207.1 [34.3 to 380.0]
  Follow-Up Visit | 18.3 [2.0 to 34.6] | 9.5 [1.5 to 21.5]

18. Secondary Outcome: Fractalkine Cytokine Levels in Urine
Description: Fractalkine Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 137.2 [8.4 to 383.8] | 58.5 [8.4 to 134.8]
  Treatment Visit | 57.0 [35.1 to 78.9] | 71.0 [48.1 to 93.9]
  Follow-Up Visit | 75.5 [20.8 to 130.2] | 86.9 [46.9 to 126.9]

19. Secondary Outcome: GRO Cytokine Levels in Urine
Description: GRO Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 13.8 [1.6 to 37.1] | 3.5 [1.6 to 7.6]
  Treatment Visit | 54.7 [8.4 to 101.0] | 224.6 [1.6 to 567.9]
  Follow-Up Visit | 28.9 [1.6 to 77.3] | 4.0 [1.6 to 9.0]

20. Secondary Outcome: IL-1RA Cytokine Levels in Urine
Description: IL-1RA Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 210.9 [1.6 to 597.4] | 44.9 [1.6 to 102.9]
  Treatment Visit | 205.2 [60.1 to 350.3] | 72.1 [35.5 to 108.7]
  Follow-Up Visit | 138.8 [1.6 to 312.3] | 64.1 [14.1 to 114.1]

21. Secondary Outcome: IL-8 Cytokine Levels in Urine
Description: IL-8 Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  Treatment Visit | 35.3 [1.6 to 79.3] | 32.9 [6.7 to 59.1]
  Follow-Up Visit | 6.3 [1.6 to 19.4] | 1.6 [1.6 to 1.6]

22. Secondary Outcome: IP-10 Cytokine Levels in Urine
Description: IP-10 Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 64.5 [1.6 to 130.7] | 23.4 [1.6 to 69.6]
  Treatment Visit | 387.8 [1.6 to 789.2] | 411.4 [1.6 to 961.1]
  Follow-Up Visit | 177.8 [1.6 to 501.8] | 23.7 [1.6 to 63.5]

23. Secondary Outcome: MCP-1 Cytokine Levels in Urine
Description: MCP-1 Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group, with MCP-1 Cytokine outcomes specified in Description.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 757.7 [1.6 to 1939.5] | 113.0 [1.6 to 263.3]
  Treatment Visit | 622.5 [1.6 to 1802.0] | 233.9 [1.6 to 494.8]
  Follow-Up Visit | 491.7 [1.6 to 1284.5] | 137.9 [83.4 to 192.4]

24. Secondary Outcome: MIP-1Beta Cytokine Levels in Urine
Description: MIP-1Beta Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 2.1 [1.6 to 3.4] | 1.6 [1.6 to 1.6]
  Treatment Visit | 16.6 [1.6 to 41.4] | 22.0 [1.6 to 66.7]
  Follow-Up Visit | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]

25. Secondary Outcome: VEGF Cytokine Levels in Urine
Description: VEGF Cytokine levels in urine collected from subjects were measured at the screening visit, during experimental infection and at the follow-up visit. Only cytokines detected during the treatment visit upon experimental infection or day 5 in > 50% of both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of quantitation are assigned 1/2 the lower limit of quantitation for calculation of mean values; limits of 95% confidence intervals are bounded by 1/2 the lower limit of quantitation and the upper limit of quantitation for each cytokine. Only the cytokines measured in both the urine and peripheral blood samples are included. Cytokine outcome values reported below the limit of detection are excluded.
Time Frame: as for outcome 4
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25
Number analyzed (Participants) | 5 | 5
pg/mL
  Screening Visit | 104.9 [9.2 to 242.5] | 45.3 [9.2 to 106.3]
  Treatment Visit | 171.8 [9.2 to 399.6] | 111.3 [9.2 to 226.4]
  Follow-Up Visit | 185.1 [9.2 to 430.4] | 71.8 [9.2 to 171.3]

26. Secondary Outcome: Pattern of Gonococcal Gene Expression in Urine Sediment
Description: RNA-seq is the standard method for measuring bacterial gene expression.
Time Frame: Day 1 through Day 5
Population: All participants in the single-strain infection groups, consisting of the Mutant FA7527 - LptA group and Wild-type FA1090 A25 group. Samples obtained were not adequate for analysis with current testing methods
Groups:
- Mutant FA7527: Participants received a bacterial inoculum containing only the isogenic LptA mutant N. gonorrhoeae strain. Mandatory rescue therapy in a single dose, on participant request, at the onset of symptoms or on the 5th study day after inoculation.
Arm/Group | Mutant FA7527 | Wild-type FA1090 A25
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Quantity of Gonococcal Gene Expression in Urine Sediment
Description: RNA-seq is the standard method for measuring bacterial gene expression.
Time Frame: Day 1 through Day 5
Population: All participants that received bacterial inoculum. Samples obtained were not adequate for analysis with current testing methods
Arm/Group | Mutant FA7527 - LptA | Wild-type FA1090 A25 | Mixed FA7527/FA1090 A25
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs that occurred within the experimental infection trial period including inoculation and one week after the follow-up visit were reported. Events noted through a telephone call approximately 7 days after the follow-up visit to assess potential AEs were also reported.
Description: The unsolicited AEs were summarized using MedDRA 15.1. The solicited AEs were assessed using MedDRA 22.1
Groups:
- Mutant FA7527: Participants received a bacterial inoculum containing only the isogenic LptA mutant N. gonorrhoeae strain.
- Wild-type FA1090 A25: Participants received a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain.
- Mixed FA7527/FA1090 A25: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic LptA mutant and WT strain.
Arm/Group | Mutant FA7527 | Wild-type FA1090 A25 | Mixed FA7527/FA1090 A25
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 4/5 | 5/5 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mutant FA7527 (N=5) | Wild-type FA1090 A25 (N=5) | Mixed FA7527/FA1090 A25 (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Instillation Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral Discharge (Renal and urinary disorders) | 3 (3) | 5 (5) | 5 (6)
Urethritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Irritation or Itching (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04870138/Prot_SAP_000.pdf